CLINICAL TRIAL: NCT02246192
Title: Application of PRGF (Plasma Rich in Growth Factors) to Reduce the Healing Time After Pilonidal Sinus Excision. A Randomized 5-years Prospective Controlled Trial.
Brief Title: Use of Plasma Rich in Growth Factors (PRGF) in Pilonidal Sinus Excision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Quiron Sagrado Corazon (Other)
Responsible Party: Principal Investigator, Juan Bellido Luque.MD, Ph.D, Hospital Quiron Sagrado Corazon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Sinusprgf
Record Dates: First submitted 2014-08-13; First posted 2014-09-22 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Pilonidal Sinus
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (Experimental): sinus pilonidal excision and standard cares
  Interventions: Procedure: sinus pilonidal excision and standard cares
- PRGF group (Experimental): sinus pilonidal excision+ PRGF
  Interventions: Procedure: sinus pilonidal excision+ PRGF

INTERVENTIONS:
Procedure: sinus pilonidal excision+ PRGF — open sinus pilonidal excision and plasma rich grow factor infiltration intra and postoperatively
  Arms: PRGF group
Procedure: sinus pilonidal excision and standard cares — sinus pilonidal excision and postoperative standard care with povidone daily
  Arms: control group

SUMMARY:
The use of plasma rich in growth factors in wound excision pilonidal sinus could improve the healing process of the wound, when compared with the usual technique of daily local healing. The investigators propose the objective of evaluating the efficacy of intra- and postoperative application of plasma rich in growth factors, to reduce healing time and complications, arising from its removal, compared to the standard surgical treatment.

DETAILED DESCRIPTION:
prospective randomized control trial, comparing PRGF application vs daily local care(betadine +saline) in sinus pilonidal wound excision. PRGF is extracted from de patient blood and infiltrated in the pilonidal wound every week. this treatment is compared with betadine and saline wound care in terms of wound healing time, pospoperative pain and other complications.

this study try to keeps the advantages of using open technique for pilonidal desease( low recurrence rate and surgical site infections) and improving the disadvantages (high wound healing time and postperative pain with wore quality of life) when it´s compared with direct closure or flap techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients among 13 and 65 years old
* Possibility of observation during the follow-up period
* Patients who have read and signed informed consent

Exclusion Criteria:

* Abscessed pilonidal sinus
* Recurrent pilonidal sinus
* Patients treated with immunosuppressive drugs or anticoagulants

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
healing time(days) of pilonidal sinus wound excision | 6 months

SECONDARY OUTCOMES:
postoperative pain | 1 month
  using VAS to assess postoperative pain

OTHER OUTCOMES:
postoperative bleeding | 1 week
surgical site infection rate | 1 month
sinus recurrence rate | 4 years
quality of life | 6 months
  this measure is assessed asking the possibility of standing in Water closet(WC) or walking correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Bellido Luque, Principal Investigator — Quirón Sagrado Corazón Hospital, Seville, Spain